CLINICAL TRIAL: NCT01774240
Title: Incidence, Severity and Treatment of Delirium in Cardiac Surgery Patients: A Before-after Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Vibeke Lind Jørgensen, MD, PhD, resident, Rigshospitalet, Denmark
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VJ1
Record Dates: First submitted 2013-01-01; First posted 2013-01-23 (Estimated); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Delirium
Keywords: Delirium; Cardiac surgery; DOS scale
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- before (No Intervention): no systematic approach
- after (Experimental): systematic screening and treatment of delirium
  Interventions: Other: systematic screening and treatment of delirium

INTERVENTIONS:
Other: systematic screening and treatment of delirium — systematic screening for delirium with DOS scale and CAM ICU. In case of delirium, treatment according to guidelines.
  Arms: after

SUMMARY:
Delirium is a common yet under diagnosed condition in hospitalized patients, and the incidence have not previously been described in Danish cardiac surgery patients. The present study seeks to describe the incidence and duration of delirium in this group of patients, before and after the introduction of standardized screening tool and a guideline for treatment of delirium after cardiac surgery.

DETAILED DESCRIPTION:
Delirium is a common yet under diagnosed condition in cardiac surgery patients, and may cause prolonged cognitive impairment and increased risk of complications. Patients are at risk of e.g. pulling catheters and lines and may fall attempting to get out of bed. The aging patient population present with many risk factors for developing delirium, but diagnostic tools have been few. Almost 50% present with hypoactive delirium, which is often not diagnosed, nor treated correctly. To optimize effect, treatment should be initiated early, maintained until clinical improvement is observed, and then tapered gradually. Recently, Delirium Observation Screening scale (DOS scale) was developed and validated in elective cardiac surgery patients in the Netherlands, with interesting results. This encouraged us to evaluate the effects of systematic delirium screening and treatment in cardiac surgery patients. To our knowledge, no prior studies have evaluated use of DOS scale in this context.

OBJECTIVES To evaluate the incidence and severity of delirium, and the effects of standardized treatment in a population of Danish cardiac surgery patients.

ELIGIBILITY:
Inclusion Criteria:

* adult patients admitted for cardiac surgery at department of cardiothoracic surgery, Rigshospitalet, denmark

Exclusion Criteria:

* patients under age 18,
* patients that died within 24 hours after admission.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2012-04; Primary Completion 2012-10 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
number of delirium free days | 14 days
  number of delirium free days are calculated as percentage of length of stay (LOS) in days.
  Participants will be followed for the duration of hospital stay, an expected average of 2 weeks

SECONDARY OUTCOMES:
complication rates | 14 days
  complications: respiratory, re-operation, infection, acute kidney injury (AKI), cerebral, cardiac, bleeding.
  participants will be followed for the duration of hospital stay, an expected average of 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Vibeke L Jorgensen, MD, PhD, Principal Investigator — Resident
Locations (1):
- Department of cardiothoracic surgery and intensive care 4142, Rigshospitalet, Blegdamsvej 6, Copenhagen, Denmark